CLINICAL TRIAL: NCT05205655
Title: Canine Olfactory Detection and Its Relevance for the Medical Identification of Patients With COVID-19
Brief Title: Detection Dogs as a Help in the Detection of COVID-19
Acronym: COVDOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Universitaire Sahloul (Other)
Responsible Party: Principal Investigator, Riadh Boukef, PROFESSOR, Hôpital Universitaire Sahloul
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: CovDog
Record Dates: First submitted 2022-01-23; First posted 2022-01-25 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
Keywords: Biomedical detection dogs; Olfaction; Olfactory sense; Screening method; Sniffer dogs
MeSH Terms: conditions — COVID-19; Anosmia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- positive group (Active Comparator): asymptomatic or mildly symptomatic participants positive for SARS-CoV-2 RNA
  Interventions: Behavioral: collection of odour samples
- negative group (Experimental): no evidence of SARS-CoV-2 by real-time RT-PCR
  Interventions: Behavioral: collection of odour samples

INTERVENTIONS:
Behavioral: collection of odour samples — Odours will be collected by participants by putting sterile compresses under the armpits for at least 4 h.

SUMMARY:
Canine olfactive detection has proven its efficacy in numerous situations (explosives, drugs, bank notes…) including for early diagnosis of human diseases: various cancers, alert of diabetic or epileptic people in immediate alarm of crisis.

DETAILED DESCRIPTION:
Fighting such a viral outbreak requires a widespread testing, one of the key measures for tackling the pandemic. In June 2020, facing a decline of COVID-19, it is possible to say that countries that have mastered their outbreak, and were able to maintain the number of infected people low, need to perform fewer test to correctly monitor the outbreak, than those countries where the virus has spread more widely. And for the same reasons, the timing of testing is also crucial. A high rate of testing will be way more effective to slow an outbreak if conducted earlier on, at a time when there is fewer infectious

The aim of this study is to evaluate if the sweat produced by COVID-19 persons (SARS-CoV-2 PCR positive) has a different odour for trained detection dogs than the sweat produced by non COVID-19 persons. The study was conducted on 3 sites, following the same protocol procedures, and involved a total of 18 dogs. A total of 198 armpits sweat samples were obtained from different hospitals. For each involved dog, the acquisition of the specific odour of COVID-19 sweat samples required from one to four hours, with an amount of positive samples sniffing ranging from four to ten.

ELIGIBILITY:
Inclusion Criteria:

* Due to have a coronavirus swab test in the previous 24 hours
* Aged ≥ 18 years
* Suspected mild COVID-19 symptoms or have been exposed to COVID-19
* Written informed consent provided

Exclusion Criteria:

* Aged < 18 years
* Written informed consent not provided
* Unable or unwilling to put a compresses for at least 4 h

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity precision of dogs to detect people with COVID-19 by their odour. | 1 months
  The main study is designed to measure the sensitivity and specificity of the dogs to detect participants infected with SARS-CoV-2. Dogs will be trained in K9 dog center for a period of 6-8 weeks to give a behavior response to positive samples. During training the reaction of each dog to a positive sample will be observed (i.e. standing, sitting or lying down) and this indicating behaviour reinforced by rewarding the dog. The dog's diagnostic accuracy will then be determined in a double-blinded study. Here the trainer and technician using the computer to record the results of the study are blinded to the identity of each sample until the trainer calls the final decision (positive or negative) based on the response of the dog to the sample.

CONTACTS AND LOCATIONS:
Overall Officials: Riadh Boukef, professor, Principal Investigator — CHU Sahloul, Sousse, Tunisia
Locations (1):
- Riadh Boukef, Sahloul, Sousse Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No